CLINICAL TRIAL: NCT00569712
Title: A Pilot Comparative Study of the Genomic Molecular and Clinical Profiles of Patients With Lung Cancer, COPD, or Asthma Treated With Symbicort Turbuhaler
Brief Title: Studying Genes in Blood and Lung Fluid Samples From Patients With Chronic Obstructive Pulmonary Disease With or Without a Previous Diagnosis of Lung Cancer or With Asthma Treated With Budesonide and Formoterol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000577434; BCCA-H06-00209; ZENECA-BCCA-H06-00209
Record Dates: First submitted 2007-12-06; First posted 2007-12-07 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Lung Cancer; Precancerous Condition
Keywords: non-small cell lung cancer; precancerous condition
MeSH Terms: conditions — Lung Neoplasms; Precancerous Conditions; Carcinoma, Non-Small-Cell Lung | interventions — Budesonide; DNA Methylation; Comparative Genomic Hybridization; Microarray Analysis; Bronchoalveolar Lavage; Immunoenzyme Techniques; Bronchoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: budesonide/formoterol fumarate dihydrate inhalation aerosol
Genetic: DNA methylation analysis
Genetic: comparative genomic hybridization
Genetic: microarray analysis
Other: bronchoalveolar lavage
Other: immunoenzyme technique
Other: laboratory biomarker analysis
Procedure: bronchoscopy

SUMMARY:
RATIONALE: Studying the genes expressed in samples of blood and lung fluid in the laboratory from patients receiving budesonide and formoterol may help doctors learn more about the effect of budesonide and formoterol on gene expression and biomarkers.

PURPOSE: This clinical trial is studying genes in blood and lung fluid samples from patients with chronic obstructive pulmonary disease, with or without a previous diagnosis of lung cancer, or with asthma treated with budesonide and formoterol.

DETAILED DESCRIPTION:
OBJECTIVES:

* To collect and integrate background information on the genetic, epigenetic, and gene expression profiles of small airway cells and markers of inflammation in bronchoalveolar lavage fluid and blood from patients with chronic obstructive pulmonary disease (COPD) with or without a prior diagnosis of lung cancer and from patients with asthma.
* To examine the effects of budesonide/formoterol fumarate dihydrate inhalation aerosol (Symbicort Turbuhaler) on methylation and gene expression profiles of airway cells as well as on inflammatory, oxidant, and other pathways in these patients.
* To determine if it would be feasible to conduct a larger study that would allow a definitive analysis of the differences in the bronchial cells and the inflammatory proteins in bronchial secretions and blood from patients with COPD with or without a prior diagnosis of lung cancer.

OUTLINE: Patients receive budesonide/formoterol fumarate dihydrate inhalation aerosol (Symbicort Turbuhaler) twice daily for 4 weeks in the absence of disease progression or unacceptable toxicities.

Patients undergo blood sample collection and bronchoscopy at baseline and at 4 weeks. Blood and bronchoalveolar fluid samples are analyzed for inflammatory biomarker measurements. Bronchial brushing cell samples are analyzed by comparative genomic hybridization array, whole genome methylation array, and gene expression profiling.

After completion of study treatment, patients are followed at 1 week by telephone interview.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Former smoker with a 30 pack-year smoking history and mild to moderate degree of airflow obstruction, meeting the following criterion:

    * GOLD class 1 or 2 chronic obstructive pulmonary disease (COPD), defined as a post-bronchodilator FEV_1 < 80% of predicted and FEV_1 to FVC ratio < 70%
  * Former smoker with COPD and has undergone a prior curative resection for stage 0 or I non-small cell lung cancer
  * Non-smoker with mild to moderate bronchial asthma not already on inhaled corticosteroids, meeting the following criterion:

    * Fully reversible airflow obstruction and post-bronchodilator FEV_1 > 80% of predicted
* No invasive cancer on bronchoscopy or abnormal spiral chest CT scan suspicious of lung cancer

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Not pregnant or nursing
* Fertile patients must use effective contraception
* Willing to use study drug twice daily regularly
* Willing to undergo a bronchoscopy
* Not planning to donate blood during study participation
* No known or suspected hypersensitivity to budesonide, formoterol fumarate dihydrate, or excipients in study drug
* No known reaction to xylocaine
* No history of allergy to Symbicort, Pulmicort, or Oxeze Turbuhaler
* No significant medical condition, such as acute or chronic respiratory failure, unstable angina, uncontrolled congestive heart failure, or bleeding disorder that, in the opinion of the investigator, may either put the patient at risk due to study participation or preclude the patient's ability to complete the study
* No travel or planned hospitalization that would preclude the patient's ability to complete the study

PRIOR CONCURRENT THERAPY:

* More than 6 months since prior and no other concurrent inhaled corticosteroids (e.g., budesonide [Pulmicort Turbuhaler], fluticasone [Flovent], beclomethasone dipropionate [QVAR], or fluticasone/salmeterol [Advair])
* More than 6 months since prior and no concurrent oral steroids (e.g., prednisone)
* No concurrent montelukast
* No concurrent immunomodulatory or immunosuppressive medication (e.g., anti-TNF or methotrexate)
* No concurrent beta-adrenergic blockers (e.g., atenolol or inderal), orally or as eye drops

Ages: 45 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Changes in the concentrations of cytokines in plasma and bronchoalveolar lavage fluid as well as gene expression profiles before and after treatment with budesonide/formoterol fumarate dihydrate inhalation aerosol (Symbicort Turbuhaler) | 24 months
Determination of DNA alterations in bronchial cells | 24 months
Correlation of molecular features (e.g., methylation or gene expression changes) with biological features | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Lam, MD, Principal Investigator — British Columbia Cancer Agency
Locations (1):
- British Columbia Cancer Agency - Vancouver Cancer Centre, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Um SJ, Lam S, Coxson H, Man SF, Sin DD. Budesonide/formoterol enhances the expression of pro Surfactant Protein-B in lungs of COPD patients. PLoS One. 2013 Dec 26;8(12):e83881. doi: 10.1371/journal.pone.0083881. eCollection 2013. PMID 24386300